CLINICAL TRIAL: NCT06015308
Title: A Randomized, Double-blind, Placebo-controlled Phase 2 Study to Evaluate the Effect of Amlitelimab on Vaccine Antibody Responses in Adult Participants With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Investigate Vaccine Responses in Subcutaneous Amlitelimab Treated Atopic Dermatitis Participants Aged 18 Years and Older Compared With Placebo
Acronym: HYDRO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SFY17915; U1111-1280-8357 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Dermatitis Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Amlitelimab (Experimental): Participants will receive amlitelimab and vaccines as per protocol.
  Interventions: Drug: Amlitelimab; Biological: Tdap vaccine; Biological: PPS vaccine
- Placebo (Placebo Comparator): Participants will receive placebo matching amlitelimab and vaccines as per protocol.
  Interventions: Drug: Placebo; Biological: Tdap vaccine; Biological: PPS vaccine

INTERVENTIONS:
Drug: Amlitelimab — Subcutaneous injection in abdomen, outer thigh, or upper arm
  Arms: Amlitelimab
Drug: Placebo — Subcutaneous injection in abdomen, outer thigh, or upper arm
  Arms: Placebo
Biological: Tdap vaccine — Intramuscular (IM) injection into the deltoid muscle of the upper arm
Biological: PPS vaccine — Intramuscular or subcutaneous injection into the deltoid muscle of the upper arm

SUMMARY:
This is a Phase 2, multicenter, randomized, double-blind placebo controlled, 2-arm study to evaluate the effect of amlitelimab on vaccine antibody responses, and the safety of amlitelimab concurrently administered with non-live vaccines in adult participants with moderate-to-severe atopic dermatitis (AD).

The purpose of this study is to compare the immune responses to concomitantly administered Boostrix (tetanus, diphtheria, and acellular pertussis [Tdap]) and Pneumovax 23 (PPSV) vaccines in adult participants with moderate-to-severe AD treated with amlitelimab versus placebo. The study will evaluate the percentage of participants achieving a positive anti-tetanus response at Week 16 (primary endpoint) and a positive anti-pneumococcal response at Week 16 (key secondary endpoint).

Study details include:

The study duration will be up to 36 weeks (for participants not entering the LTS17367 [RIVER-AD]).

The screening period will be 9 days to 4 weeks. The treatment duration will be up to 16 weeks. The post-treatment safety follow-up period will be16 weeks. The number of visits will be up to 7 (or 6 for those entering LTS17367 [RIVER-AD]).

DETAILED DESCRIPTION:
The study duration will be up to 36 weeks

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age (when signing informed consent form)
* Diagnosis of AD for at least 1 year (defined by the American Academy of Dermatology Consensus Criteria)
* Documented history (within 6 months before screening) of either inadequate response or inadvisability to topical treatments
* Validated Investigator Global Assessment scale for atopic dermatitis (vIGA-AD) of 3 or 4 at baseline visit
* Eczema area and severity index (EASI) score of 12 or higher at baseline
* AD involvement of 10% or more of body surface area (BSA) at baseline
* Able and willing to comply with requested study visits and procedures
* Body weight ≥40 kg and ≤150 kg

Exclusion Criteria:

* Skin co-morbidity that would adversely affect the ability to undertake AD assessments
* Receipt of any vaccine (expect influenza and COVID-19 vaccines) within 3 months prior to screening
* Receipt of any pneumococcal vaccine within approximate timeframe of 5 years prior to screening
* Prior receipt of two or more doses of Pneumovax 23 at any time
* Receipt of any tetanus-, diphtheria-, or pertussis-containing vaccine within approximate timeframe of 5 years prior to screening
* Participants for whom administration of the pneumococcal vaccine provided in this study is contraindicated or medically inadvisable, according to local label of the vaccine
* Participants for whom administration of the tetanus, diphtheria, and pertussis vaccine provided in this study is contraindicated or medically inadvisable, according to local label of the vaccine
* Having received any of the specified therapy within the specified timeframe(s) prior to the baseline visit
* Known history of or suspected significant current immunosuppression
* Any malignancies or history of malignancies prior to baseline (excluding non-melanoma skin cancer excised and cured >5 years prior to baseline)
* History of solid organ or stem cell transplant
* Any active or chronic infection including helminthic infection requiring systemic treatment within 2 weeks prior baseline
* Positive for human immunodeficiency virus (HIV), Hepatitis B or hepatitis C at screening visit
* Participants with active tuberculosis (TB), latent TB, a history of incompletely treated TB, suspected extrapulmonary TB infection, or who are at high risk of contracting TB

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2026-01-16 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with a positive tetanus response at Week 16 | Week 16
  Positive tetanus response is defined as a ≥4-fold increase from pre-vaccination at baseline in anti-tetanus immunoglobulin G [IgG] titer for participants with a pre-vaccination tetanus antibody titers ≥0.1 IU/mL or a titer of ≥0.2 IU/mL for participants with pre-vaccination titers of <0.1 IU/mL.

SECONDARY OUTCOMES:
Percentage of participants with a positive pneumococcal vaccine response at Week 16 | Week 16
  Positive pneumococcal vaccine response is defined as a ≥2-fold increase from baseline in anti-pneumococcal antibodies (APAb) against >50% of the 23 serotypes.
Percentage of participants who experienced treatment-emergent adverse events (TEAE), including serious adverse events (SAE) and adverse events of special interest (AESI) | Week 0 up to Week 32
Percentage of participants with potentially clinically significant abnormalities (PCSA) for vital signs and clinical laboratory assessments | Week 0 up to Week 32
Percentage of participants discontinued from study treatment due to TEAEs | Week 0 up to Week 32
Proportion of participants with validated Investigator Global Assessment scale for atopic dermatitis (vIGA-AD) of 0 (clear) or 1 (almost clear) and a reduction of ≥2 points from baseline at Week 16 | Week 16
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Proportion of participants with a ≥75% reduction in EASI score (EASI-75) from baseline at Week 16 | Week 16
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD using a 4-point scale; 0 (absent) to 3 (severe).
Serum amlitelimab concentrations | Week 0 up to Week 16
Incidence of antidrug antibodies (ADAs) of amlitelimab | Week 0 up to Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (57):
- United States (47):
  - Clinical Research Center of Alabama - Homewood- Site Number : 8401101, Birmingham, Alabama
  - Center for Dermatology and Plastic Surgery- Site Number : 8401119, Scottsdale, Arizona
  - Orange County Clinical Trials- Site Number : 8401271, Anaheim, California
  - First OC Dermatology- Site Number : 8401025, Fountain Valley, California
  - Center for Dermatology Clinical Research- Site Number : 8401018, Fremont, California
  - Valley Research- Site Number : 8401097, Fresno, California
  - Paradigm Clinical Research Centers- Site Number : 8401273, La Mesa, California
  - Sunwise Clinical Research- Site Number : 8401022, Lafayette, California
  - Antelope Valley Clinical Trials- Site Number : 8401099, Lancaster, California
  - Torrance Clinical Research- Site Number : 8401027, Lomita, California
  - Clinical Science Institute- Site Number : 8401028, Santa Monica, California
  - Velocity Clinical Research - Denver Site Number : 8401168, Denver, Colorado
  - Daxia Trials- Site Number : 8401145, Boca Raton, Florida
  - Encore Medical Research of Boynton Beach- Site Number : 8401030, Boynton Beach, Florida
  - Alliance for Multispeciality Research - Fort Myers- Site Number : 8401111, Fort Myers, Florida
  - Doral Medical Research- Site Number : 8401094, Hialeah, Florida
  - C&R Research Services - Kendall- Site Number : 8401029, Kendall, Florida
  - Acevedo Clinical Research Associates- Site Number : 8401088, Miami, Florida
  - Future Care Solution - Miami- Site Number : 8401144, Miami, Florida
  - Sanchez Clinical Research- Site Number : 8401095, Miami, Florida
  - Florida International Research Center- Site Number : 8401091, Miami, Florida
  - Wellness Clinical Research - Miami Lakes- Site Number : 8401109, Miami Lakes, Florida
  - K2 South Orlando - South Orange Avenue- Site Number : 8401268, Orlando, Florida
  - SEC Clinical Research- Site Number : 8401270, Pensacola, Florida
  - Global Clinical Professionals (GCP)- Site Number : 8401045, St. Petersburg, Florida
  - Clinical Research Trials of Florida- Site Number : 8401023, Tampa, Florida
  - Paradigm Clinical Research - Boise- Site Number : 8401272, Boise, Idaho
  - Skin Sciences- Site Number : 8401039, Louisville, Kentucky
  - Velocity Clinical Research at The Dermatology Clinic- Site Number : 8401072, Baton Rouge, Louisiana
  - BRCR Global Gretna- Site Number : 8401243, Gretna, Louisiana
  - Boeson Research - Missoula- Site Number : 8401269, Missoula, Montana
  - Henderson Clinical Trials- Site Number : 8401169, Henderson, Nevada
  - Skin Search Rochester- Site Number : 8401216, Rochester, New York
  - Velocity Clinical Research - Durham- Site Number : 8401175, Durham, North Carolina
  - Velocity Clinical Research - Springdale- Site Number : 8401153, Cincinnati, Ohio
  - Velocity Clinical Research - Medford- Site Number : 8401170, Medford, Oregon
  - Vial Health - DermDox Dermatology- Site Number : 8401031, Camp Hill, Pennsylvania
  - Velocity Clinical Research - Providence- Site Number : 8401179, East Greenwich, Rhode Island
  - Velocity Clinical Research - Charleston - Ashley Town Center Drive- Site Number : 8401174, Charleston, South Carolina
  - Velocity Clinical Research - Columbia- Site Number : 8401176, Columbia, South Carolina
  - Velocity Clinical Research - Austin- Site Number : 8401173, Cedar Park, Texas
  - Modern Research Associates- Site Number : 8401093, Dallas, Texas
  - Heights Dermatology & Aesthetic Center- Site Number : 8401143, Houston, Texas
  - Dermatology Clinical Research Center of San Antonio- Site Number : 8401100, San Antonio, Texas
  - Discovery Clinical Trials - San Antonio - Stone Oak Parkway- Site Number : 8401026, San Antonio, Texas
  - Stryde Research - Epiphany Dermatology- Site Number : 8401185, Southlake, Texas
  - Ogden Clinic Mountain View (Avacare) Site Number : 8401167, Pleasant View, Utah
- Canada (10):
  - Investigational Site Number : 1240019, Calgary, Alberta
  - Investigational Site Number : 1240023, Calgary, Alberta
  - Investigational Site Number : 1240016, Edmonton, Alberta
  - Investigational Site Number : 1240014, Barrie, Ontario
  - Investigational Site Number : 1240020, Hamilton, Ontario
  - Investigational Site Number : 1240017, London, Ontario
  - Investigational Site Number : 1240018, Newmarket, Ontario
  - Investigational Site Number : 1240024, Richmond Hill, Ontario
  - Investigational Site Number : 1240021, Toronto, Ontario
  - Investigational Site Number : 1240026, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: SFY17915 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25504&tenant=MT_SNY_9011